CLINICAL TRIAL: NCT00784836
Title: A Multicenter, Open-Label, Immunogenicity and Safety Study of Avonex® (Interferon Beta-1a) 30 mcg Administered Subcutaneously to Subjects With Relapsing Multiple Sclerosis
Brief Title: Immunogenicity and Safety of Subcutaneously-administered Avonex (Interferon Beta-1a) in Multiple Sclerosis (MS) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early by Sponsor for business reasons unrelated to safety.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108MS303
Record Dates: First submitted 2008-10-29; First posted 2008-11-04 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis - Relapsing
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avonex (Experimental): Avonex 30 mcg given subcutaneously, once weekly, for 18 months.
  Interventions: Drug: BG9418 (interferon beta 1-a)

INTERVENTIONS:
Drug: BG9418 (interferon beta 1-a)
  Other Names: Avonex

SUMMARY:
The primary objective of the study was to evaluate the immunogenicity of Avonex® (interferon beta-1a) 30 mcg when administered subcutaneously (SC) to interferon-naïve participants with relapsing multiple sclerosis. The secondary objective of this study was to evaluate the safety and tolerability of Avonex® 30 mcg when administered SC to interferon-naïve subjects with relapsing MS.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Male or female aged 18- to 60-years-old, inclusive, at the time of informed consent.
* Must have a diagnosis of relapsing MS.
* Must have a screening Expanded Disability Status Scale (EDSS) score between 0 and 6.0, inclusive.
* All male subjects and female participants of child-bearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last study dose of Avonex.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions.
* Diagnosed with Primary progressive, secondary progressive, or progressive relapsing MS.
* Known allergy to any component of the Avonex formulation.
* History of any clinically significant (as determined by the investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric renal, or other major disease.
* Subjects with history of malignant disease, including solid tumors and hematologic malignancies.
* History of seizure disorder or unexplained blackouts OR history of a seizure within 3 months prior to Day 1.
* History of suicidal ideation within 3 months prior to Day 1 or an episode of severe depression within 3 months prior to Day 1. Severe depression is defined as any episode of depression that requires hospitalization, or the initiation of antidepressant therapy, or an increase in the dose of an existing regimen of antidepressant therapy.
* Clinically significant abnormal electrocardiogram (ECG) values as determined by the investigator.
* Known history of, or a positive test result for, human immunodeficiency virus (HIV).
* Known history of, or a positive test result for hepatitis C virus.
* Abnormal screening blood tests exceeding any of the limits defined below:

  1. Alanine transaminase/serum glutamate pyruvate transaminase (ALT/SGPT) greater than 2 times the upper limit of normal or aspartate transaminase/serum glutamic oxaloacetic transaminase or bilirubin.
  2. Total white blood cell count (WBC) <3700 cells/mm
  3. Platelet count <150,000 cells/mm
  4. Hemoglobin <10 g/dL in female subjects; <11 g/dL in male subjects
  5. Serum creatinine >upper limit of normal (ULN)
  6. Prothrombin time (PT) or activated partial thromboplastin time (aPTT) > 1.2*ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - MS Center at Texas Neurology, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study expected an enrollment of 150 participants, but terminated after 3 were enrolled.
Period: Overall Study
Arm/Group | Avonex
Started | 3
Completed | 0 (The study was terminated early by the Sponsor for business reason not related to safety.)
Not Completed | 3
Not completed — Early Study Termination | 3

BASELINE CHARACTERISTICS:
Arm/Group | Avonex
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 60 years | 3
  > 60 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Neutralizing Antibodies (NAbs) to Interferon-beta (IFN-beta)
Description: The presence of antibodies to IFN-beta in human serum, determined using a tiered approach involving a screening Enzyme-Linked ImmunoSorbent Assay (ELISA) to detect binding antibodies (BAbs). Positive samples characterized and titrated in a cell-based neutralizing antibody (NAb) assay.
Time Frame: assessed every 3 months up to 18 months
Population: The study was terminated early before any of the 3 enrolled subjects completed the study; therefore, no statistical analysis was performed.
Arm/Group | Avonex
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Planned for up to 18 months plus 30 days; actual study duration was 111 days.
Measure: Number; unit: participants
Arm/Group | Avonex
Number analyzed (Participants) | 3
participants
  AEs | 3
  SAEs | 0

ADVERSE EVENTS:
Time Frame: Planned for up to 18 months plus 30 days; actual study duration was 111 days.
Arm/Group | Avonex
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avonex (N=3)
Injection site reaction (General disorders) | 1
Influenza like illness (General disorders) | 2
Hepatic enzyme increased (Investigations) | 1

LIMITATIONS AND CAVEATS:
Early termination with partial data from 3 subjects, therefore, no statistical analysis performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.